CLINICAL TRIAL: NCT04682119
Title: A Safety, Tolerability and Pharmacokinetic Study of Single and Multiple Doses of LY3526318 in Healthy Participants
Brief Title: A Safety Study of LY3526318 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 17807; 2020-004290-46 (EudraCT Number); J2D-MC-CVAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2020-12-22; First posted 2020-12-23 (Actual); Results first posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LY3526318 (Part A) (Experimental): 250 mg, 100 milligram (mg) LY3526318 administered orally as single ascending doses under fasted or fed condition.
  Interventions: Drug: LY3526318
- LY3526318 (Part B) (Experimental): 250 mg LY3526318 administered orally as multiple doses under fasted or fed condition.
  Interventions: Drug: LY3526318
- Placebo (Part A) (Placebo Comparator): Placebo administered orally under fasted or fed condition.
  Interventions: Drug: Placebo
- Placebo (Part B) (Placebo Comparator): Placebo administered orally under fasted or fed condition.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3526318 — Administered orally.
  Arms: LY3526318 (Part A); LY3526318 (Part B)
Drug: Placebo — Administered orally.
  Arms: Placebo (Part A); Placebo (Part B)

SUMMARY:
The main purpose of this study is to learn more about how the drug is absorbed in to the blood stream and how it is eliminated from the body. The safety and tolerability of LY3526318 will also be evaluated when given by mouth either by single or multiple doses to healthy participants. The study will have two parts. Each participant will enroll in only one part. For each participant, Part A will last up to 44 days and Part B will last up to 50 days, including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females, as determined through medical history and physical examination
* Have a body mass index (BMI) between 18 and 32 kilograms per square meter (kg/m²)
* Have clinical laboratory test results within normal reference range

Exclusion Criteria:

* Have a history or presence of medical illness including, but not limited to, cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, convulsions, or any clinically significant laboratory abnormality
* Have an abnormality in the 12-lead electrocardiogram (ECG)
* Have a history of clinically significant multiple or severe drug allergies
* Show evidence of human immunodeficiency virus (HIV) and/or positive human HIV antibodies, hepatitis C and/or positive hepatitis C antibody, or hepatitis B and/or positive hepatitis B surface antigen.
* Have an abnormal blood pressure
* Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer)
* Are unwilling to stop herbal supplements, over the counter or prescription medicines
* Are currently enrolled in a clinical drug study or any other type of medical research judged not to be scientifically or medically compatible with this study.
* Participants with a history of drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-12-29 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study consists of 2 parts:
  * Part A: Single-ascending dose (SAD, [including a food effect (FE)]).
  * Part B: Multiple-ascending dose (MAD), [including a food effect (FE)]).
  Both parts were randomized, double-blind, and placebo-controlled.
Groups:
- Part A SAD: P1-L2-L3-L4: P1: Participants received placebo administered orally under fasted condition during period 1.
  L2: Participants received 250 milligram (mg) LY3526318 administered orally under fasted condition during period 2.
  L3: Participants received 250 mg LY3526318 administered orally in fed state after a light breakfast during period 3.
  L4: Participants received 250 mg LY3526318 administered orally in fed state after a high-fat breakfast during period 4.
- Part A SAD: L1-P1-L3-L4: L1: Participants received 100 mg LY3526318 administered orally under fasted condition during period 1.
  P1: Participants received placebo administered orally under fasted condition during period 2.
  L3: Participants received 250 mg LY3526318 administered orally in fed state after a light breakfast during period 3.
  L4: Participants received 250 mg LY3526318 administered orally in fed state after a high-fat breakfast during period 4.
- Part A SAD: L1-L2-P3-L4: L1: Participants received 100 mg LY3526318 administered orally under fasted condition during period 1.
  L2: Participants received 250 mg LY3526318 administered orally under fasted conditions during period 2.
  P3: Participants received placebo administered orally in fed state after a light breakfast during period 3.
  L4: Participants received 250 mg LY3526318 administered orally in fed state after a high-fat breakfast during period 4.
- Part A SAD: L1-L2-L3-P4: L1: Participants received 100 mg LY3526318 administered orally under fasted condition during period 1.
  L2: Participants received 250 mg LY3526318 administered orally under fasted condition during period 2.
  L3: Participants received 250 mg LY3526318 administered orally in fed state after a light breakfast during period 3.
  P4: Participants received placebo administered orally in fed state after a high-fat breakfast during period 4.
- Part B MAD: Placebo: Participants received placebo administered orally under fasted conditions on Day 1 and Day 5 and in fed state after participants ate a standard breakfast without respect to dosing time on Day 2 to Day 4.
- Part B MAD: 250 mg LY3526318: Participants received 250 mg LY3526318 administered orally under fasted conditions on Day 1 and Day 5 and in fed state after participants ate a standard breakfast without respect to dosing time on Day 2 to Day 4.
Period: Period 1
Arm/Group | Part A SAD: P1-L2-L3-L4 | Part A SAD: L1-P1-L3-L4 | Part A SAD: L1-L2-P3-L4 | Part A SAD: L1-L2-L3-P4 | Part B MAD: Placebo | Part B MAD: 250 mg LY3526318
Started | 2 | 2 | 2 | 2 | 2 | 6
All Participants Who Received at Least One Dose of Study Drug | 2 | 2 | 2 | 2 | 2 | 6
Completed | 2 | 2 | 2 | 2 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Part A SAD: P1-L2-L3-L4 | Part A SAD: L1-P1-L3-L4 | Part A SAD: L1-L2-P3-L4 | Part A SAD: L1-L2-L3-P4 | Part B MAD: Placebo | Part B MAD: 250 mg LY3526318
Started | 2 | 2 | 2 | 2 | 0 (The length of time for Part B MAD part of the study was 1 period.) | 0 (The length of time for Part B MAD part of the study was 1 period.)
Completed | 2 | 2 | 2 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Part A SAD: P1-L2-L3-L4 | Part A SAD: L1-P1-L3-L4 | Part A SAD: L1-L2-P3-L4 | Part A SAD: L1-L2-L3-P4 | Part B MAD: Placebo | Part B MAD: 250 mg LY3526318
Started | 2 | 2 | 2 | 2 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Part A SAD: P1-L2-L3-L4 | Part A SAD: L1-P1-L3-L4 | Part A SAD: L1-L2-P3-L4 | Part A SAD: L1-L2-L3-P4 | Part B MAD: Placebo | Part B MAD: 250 mg LY3526318
Started | 2 | 2 | 2 | 2 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Part A SAD: Sequence P1-L2-L3-L4: P1: Participants received placebo administered orally under fasted condition during period 1.
  L2: Participants received 250 mg LY3526318 administered orally under fasted condition during period 2.
  L3: Participants received 250 mg LY3526318 administered orally in fed state after a light breakfast during period 3.
  L4: Participants received 250 mg LY3526318 administered orally in fed state after a high-fat breakfast during period 4.
- Part A: L1-L2-L3-P4: L1: Participants received 100 mg LY3526318 administered orally under fasted condition during period 1 L2: Participants received 250 mg LY3526318 administered orally under fasted condition during period 2.
  L3: Participants received 250 mg LY3526318 administered orally in fed state after a light breakfast during period 3.
  P4: Participants received placebo administered orally in fed state after a high-fat breakfast during period 4.
- Total: Total of all reporting groups
Arm/Group | Part A SAD: Sequence P1-L2-L3-L4 | Part A SAD: L1-P1-L3-L4 | Part A SAD: L1-L2-P3-L4 | Part A: L1-L2-L3-P4 | Part B MAD: Placebo | Part B MAD: 250 mg LY3526318 | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (4) | 31 (11) | 59 (3) | 43 (13) | 31 (14) | 35 (21) | 40 (16.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 2 | 4 | 10
  Male | 1 | 1 | 1 | 1 | 0 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 2 | 2 | 1 | 2 | 2 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 1 | 2 | 1 | 6 | 13
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Netherlands | 2 | 2 | 2 | 2 | 2 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Part A - SAD, Pharmacokinetics (PK): Area Under the Concentration Time Curve From Time 0 to Infinity (AUC 0-∞) of LY3526318
Description: Area Under the Concentration Time Curve From Time 0 to Infinity (AUC 0-∞) of LY3526318
Time Frame: Predose,1, 2, 4, 6, 8,12, 24, 48, 72, 96 hours post-dose
Population: Part A - SAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Groups:
- Part A - SAD: 250 mg LY3526318 Fed (Light Breakfast): Participants received 250 mg LY3526318 administered orally in fed state after a light breakfast.
- Part A - SAD: 250 mg LY3526318 Fed (High Fat Meal): Participants received 250 mg LY3526318 administered orally in fed state after a high-fat breakfast.
- Part A - SAD: 250 mg LY3526318 Fasted: Participants received 250 mg LY3526318 administered orally under fasted condition.
- Part A - SAD: 100 mg LY3526318 Fasted: Participants received 100 mg LY3526318 administered orally under fasted condition.
Arm/Group | Part A - SAD: 250 mg LY3526318 Fed (Light Breakfast) | Part A - SAD: 250 mg LY3526318 Fed (High Fat Meal) | Part A - SAD: 250 mg LY3526318 Fasted | Part A - SAD: 100 mg LY3526318 Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanograms*hours per milliliter (ng*h/mL) | 147978 (37.5) | 131271 (61.8) | 137814 (58.6) | 76902 (56.1)

2. Primary Outcome: Part A - SAD, PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Description: Part A - SAD, PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Time Frame: Predose,1, 2, 4, 6, 8,12, 24, 48, 72, 96 hours post-dose
Population: Part A - SAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Part A - SAD: 250 mg LY3526318 Fed (Light Breakfast) | Part A - SAD: 250 mg LY3526318 Fed (High Fat Meal) | Part A - SAD: 250 mg LY3526318 Fasted | Part A - SAD: 100 mg LY3526318 Fasted
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 12406 (26.4) | 6199 (61.4) | 9544 (26.8) | 5441 (49.9)

3. Primary Outcome: Part B - MAD, PK: Area Under the Concentration Time Curve From Time Zero to the End of the Dosing Interval, Tau (AUC[0-tau ]) of LY3526318
Description: Part B - MAD, PK: Area Under the Concentration Time Curve From Time Zero to the End of the Dosing Interval, Tau (AUC[0-tau ]) of LY3526318
Time Frame: Day 5: Predose,1, 2, 4, 6, 8,12, 24 hours post dose
Population: Part B - MAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- Part B MAD:250 mg LY3526318: Participants received 250 mg LY3526318 administered orally under fasted conditions on Day 1 and Day 5 and in fed state after participants ate a standard breakfast without respect to dosing time on Day 2 to Day 4.
Arm/Group | Part B MAD:250 mg LY3526318
Number analyzed (Participants) | 6
ng*h/mL | 89614 (19.7)

4. Primary Outcome: Part B - MAD, PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Description: Part B - MAD, PK: Maximum Observed Drug Concentration (Cmax) of LY3526318
Time Frame: Day 5: Predose,1, 2, 4, 6, 8,12, 24 hours post dose
Population: Part B - MAD: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- Part B MAD:250 mg LY3526318 LY3526318 QD: Participants received 250 mg LY3526318 administered orally under fasted conditions on Day 1 and Day 5 and in fed state after participants ate a standard breakfast without respect to dosing time on Day 2 to Day 4.
Arm/Group | Part B MAD:250 mg LY3526318 LY3526318 QD
Number analyzed (Participants) | 6
nanograms per milliliter (ng/mL) | 10717 (35.1)

5. Secondary Outcome: Part A, SAD: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: A TEAE started on or after the date and time of the first dose of study drug administered in this study, or started prior to the study drug administration but worsened after the study drug started. Clinically significant events were defined as SAEs and other non-serious adverse events (AEs). A summary of SAEs and other non-serious AEs is located in the Reported Adverse Events module.
Time Frame: Single oral dose to up to 11 days of follow-up
Population: Part A, SAD: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Part A - SAD: Placebo Fasted: Participants received placebo administered orally under fasted condition.
- Part A - SAD: Placebo Fed (Light Breakfast): Participants received placebo administered orally in fed state after a light breakfast.
- Part A - SAD: Placebo Fed (High Fat Meal): Participants received placebo administered orally in fed state after a high-fat breakfast.
Arm/Group | Part A - SAD: Placebo Fasted | Part A - SAD: Placebo Fed (Light Breakfast) | Part A - SAD: Placebo Fed (High Fat Meal) | Part A - SAD: 100 mg LY3526318 Fasted | Part A - SAD: 250 mg LY3526318 Fasted | Part A - SAD: 250 mg LY3526318 Fed (Light Breakfast) | Part A - SAD: 250 mg LY3526318 Fed (High Fat Meal)
Number analyzed (Participants) | 4 | 2 | 2 | 6 | 6 | 6 | 6
Participants
  TEAEs | 2 | 1 | 1 | 2 | 2 | 4 | 1
  SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Part B, MAD: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: as for outcome 5
Time Frame: Up to 14 days following first dose
Population: Part B, MAD: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B MAD: Placebo | Part B MAD:250 mg LY3526318 LY3526318 QD
Number analyzed (Participants) | 2 | 6
Participants
  TEAEs | 1 | 4
  SAEs | 0 | 0

7. Secondary Outcome: Part A, Effect of a Meal on Pharmacokinetics of LY3526318: Maximum Concentration (Cmax)
Description: Part A, Effect of a meal on pharmacokinetics of LY3526318: Maximum Concentration (Cmax)
Time Frame: Predose,1, 2, 4, 6, 8,12, 24, 48, 72, 96 hours post-dose
Population: Part A, SAD: All participants who received 250 mg LY3526318 and had evaluable PK data.
Measure: Number (90% Confidence Interval); unit: unitless
Groups:
- Part A: 250 mg LY3526318: Participants received 250 mg LY3526318 administered orally in fasted state, in fed state after a light breakfast or in fed state after a high-fat breakfast.
Arm/Group | Part A: 250 mg LY3526318
Number analyzed (Participants) | 8
unitless
  Ratio of Fed Light Breakfast/ Fasted | 1.2768 [0.9030 to 1.8052]
  Ratio of Fed High Fat Meal/ Fasted | 0.6195 [0.4381 to 0.8759]

8. Secondary Outcome: Part A, Effect of a Meal on Pharmacokinetics of LY3526318: Area Under the Concentration Time Curve From Time 0 to Infinity (AUC 0-∞)
Description: Part A, Effect of a meal on pharmacokinetics of LY3526318: Area under the concentration time curve from time 0 to infinity (AUC 0-∞)
Time Frame: Predose,1, 2, 4, 6, 8,12, 24, 48, 72, 96 hours post-dose
Population: Part A, SAD: All participants who received 250 mg LY3526318 and had evaluable PK data.
Measure: Number (90% Confidence Interval); unit: unitless
Arm/Group | Part A: 250 mg LY3526318
Number analyzed (Participants) | 8
unitless
  Ratio of Fed Light Breakfast/ Fasted | 1.1341 [0.9722 to 1.3229]
  Ratio of Fed High Fat Meal/ Fasted | 0.8454 [0.7248 to 0.9862]

9. Secondary Outcome: Part A, Effect of a Meal on Pharmacokinetics of LY3526318: Time at Maximal Concentration (Tmax)
Description: Part A, Effect of a Meal on Pharmacokinetics of LY3526318: Time at Maximal Concentration (Tmax)
Time Frame: Predose,1, 2, 4, 6, 8,12, 24, 48, 72, 96 hours post-dose
Population: Part A, SAD: All participants who received 250 mg LY3526318 and had evaluable PK data
Measure: Number (90% Confidence Interval); unit: hours
Arm/Group | Part A: 250 mg LY3526318
Number analyzed (Participants) | 8
hours
  Fed Light Breakfast - Fasted | 0.00 [0.00 to 2.00]
  Fed High Fat Meal - Fasted | 0.03 [0.00 to 2.03]

ADVERSE EVENTS:
Time Frame: Baseline Up To 14 Days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Part A - SAD: Placebo Fed (Light Breakfast) | Part A - SAD: Placebo Fed (High Fat Meal) | Part A - SAD: Placebo Fasted | Part A - SAD: 250 mg LY3526318 Fed (Light Breakfast) | Part A - SAD: 250 mg LY3526318 Fed (High Fat Meal) | Part A - SAD: 250 mg LY3526318 Fasted | Part A - SAD: 100 mg LY3526318 Fasted | Part B MAD: Placebo | Part B MAD:250 mg LY3526318
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/4 | 0/6 | 0/6 | 0/6 | 0/6 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 2/4 | 4/6 | 1/6 | 2/6 | 2/6 | 1/2 | 4/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A - SAD: Placebo Fed (Light Breakfast) (N=2) | Part A - SAD: Placebo Fed (High Fat Meal) (N=2) | Part A - SAD: Placebo Fasted (N=4) | Part A - SAD: 250 mg LY3526318 Fed (Light Breakfast) (N=6) | Part A - SAD: 250 mg LY3526318 Fed (High Fat Meal) (N=6) | Part A - SAD: 250 mg LY3526318 Fasted (N=6) | Part A - SAD: 100 mg LY3526318 Fasted (N=6) | Part B MAD: Placebo (N=2) | Part B MAD:250 mg LY3526318 (N=6)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/19/NCT04682119/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/19/NCT04682119/SAP_001.pdf